CLINICAL TRIAL: NCT04275284
Title: Evaluation of Persistence of Immunogenicity Following an Open-labelled, Randomized Controlled Trial Evaluating Non-inferiority of 1+1 Compared to 2+1 Dosing Schedules of 10-valent and 13-valent Pneumococcal Conjugate Vaccine in South Africa
Brief Title: Persistence of Immunogenicity Following Reduced PCV Dosing Schedules in South African Children
Acronym: PCV1+1_FU
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Farzanah Laher, Dr, University of Witwatersrand, South Africa
Other Study IDs: PCV1+1 follow-up
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pneumonia; Meningitis
MeSH Terms: conditions — Pneumonia; Meningitis | interventions — 10-valent pneumococcal conjugate vaccine; PHiD-CV vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and nasopharyngeal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- PCV10 1+1, 6 weeks & 9 months: Follow-up of children who were previously randomized to PCV10 (Synflorix 0.5ml injection) administered at 6 weeks and 9 months of age.
  Interventions: Biological: PCV10
- PCV13 1+1, 6 weeks & 9 months: Follow-up of children who were previously randomized to PCV13 (Prevnar 13, 0.5ml injection) administered at 6 weeks and 9 months of age.
  Interventions: Biological: PCV13
- PCV10 1+1, 14 weeks & 9 months: Follow-up of children who were previously randomized to PCV10 (Synflorix 0.5ml injection) administered at 14 weeks and 9 months of age.
  Interventions: Biological: PCV10
- PCV13 1+1, 14 weeks & 9 months: Follow-up of children who were previously randomized to PCV13 (Prevnar 13, 0.5ml injection) administered at 14 weeks and 9 months of age.
  Interventions: Biological: PCV13
- PCV10 2+1, 6&14 weeks & 9 months: Follow-up of children who were previously randomized to PCV10 (Synflorix 0.5ml injection) administered at 6 weeks, 14 weeks and 9 months of age.
  Interventions: Biological: PCV10
- PCV13 2+1, 6&14 weeks & 9 months: Follow-up of children who were previously randomized to PCV13 (Prevnar 13, 0.5ml injection) administered at 6 weeks, 14 weeks and 9 months of age.
  Interventions: Biological: PCV13

INTERVENTIONS:
Biological: PCV10 — 0.5 ml injection
  Other Names: Synflorix
  Groups: PCV10 1+1, 14 weeks & 9 months; PCV10 1+1, 6 weeks & 9 months; PCV10 2+1, 6&14 weeks & 9 months
Biological: PCV13 — 0.5 ml injection
  Other Names: Prevnar13
  Groups: PCV13 1+1, 14 weeks & 9 months; PCV13 1+1, 6 weeks & 9 months; PCV13 2+1, 6&14 weeks & 9 months

SUMMARY:
This study will evaluate the persistence of immunogenicity following a reduced dosing schedule of 10- or 13-valent Pneumococcal Conjugate Vaccine (PCV10, PCV13). This is the follow-up of a randomized controlled trial in which children received a single priming dose of PCV10 or PCV13 (at 6 or 14 weeks of age) followed by booster dose at 9 months of age (1+1 schedule), compared to a 2+1 PCV schedule (6, 14 weeks of age and 9 months of age).

DETAILED DESCRIPTION:
Between 2017 and 2019, we conducted an open-labelled, randomized controlled trial to evaluate for non-inferiority in the post-booster serotype-specific geometric mean concentrations (GMC's) in children randomized to receive either PCV10 or PCV13 as a 1+1 schedule (with the first dose occurring either at 6 or 14 weeks of age) compared to infants who received a two dose primary series (6 and 14 weeks of age). All six study groups received a booster dose at 40 weeks of age, and serotype-specific IgG and opsonophagocytic activity was measured one-month post booster. Subjects were planned to be followed-up until 18 months of age as part of the initial study. In the present study, we propose to extent the follow-up of the cohort to include annual visit at 3, 4 and 5 years of age, to evaluate the sustainability of the humoral immune response of the different PCV dosing schedules.

ELIGIBILITY:
Inclusion Criteria:

1. Children between and including the ages of 36 - 38 months of age at the time of first blood sampling;
2. Subjects who previously participated in the PCV1+1 study and received the full study vaccination regime as per protocol;
3. The parent or legal guardian of the child must be able and willing to provide written informed consent for all 3 visits and comply with all study requirements;
4. The parent or legal guardian of the child must indicate the intention to remain in the study area for the duration of the trial - or be willing to bring the child for all visits.

Exclusion Criteria:

1. Receipt of any additional pneumococcal vaccine since the end of participation in the PCV1+1 study;
2. Any known or suspected immunodeficiency condition which could affect immune response to vaccination, including living with HIV;
3. Receipt of any immunoglobulins and/or blood products less than 6 months prior to blood sampling;
4. Parent/legal guardian unable or unwilling to attend scheduled study visits.

Ages: 3 Years to 5 Years | Sex: All
Age Groups: Child
Study Population: All participants who completed the PCV1+1 study and received all vaccines as specified per study protocol will be contacted to participate.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Serotype specific geometric mean antibody concentrations (GMC) | 3, 4 and 5 years of age
  To evaluate persistence of vaccine-serotype specific GMCs at 3, 4 and 5 years of age between children receiving differing 1+1 dosing schedules compared to the 2+1 dosing schedule of the same vaccine formulation (i.e. PCV10 or PCV13).

SECONDARY OUTCOMES:
Modified threshold of protection | 3, 4 and 5 years of age
  To evaluate persistence of vaccine-serotype specific serum IgG antibody concentration above the WHO-defined putative threshold for protection (≥0.35 µg/mL) and the modified serotype-specific correlate of protection against IPD as proposed by Andrews et al.(17) at 3, 4 and 5 years of between children with differing 1+1 dosing schedules compared to the 2+1 dosing schedule of the same vaccine formulation
Comparison between 6-week and 14-week primary dose | 3, 4 and 5 years of age
  To evaluate persistence of vaccine-serotype specific serum IgG antibody concentration above the WHO-defined putative threshold for protection (≥0.35 µg/mL), the modified serotype-specific correlate of protection against IPD as proposed by Andrews et al. (17) and GMC's at 3, 4 and 5 years in children receiving the 1+1 dosing schedule at either 6 weeks of age compared to those who received it at 14 weeks of age, stratified for the individual vaccine formulation (PCV10 and PCV13).
Colonization outcome | 3, 4 and 5 years of age
  To compare the prevalence of vaccine-serotype (stratified by PCV10 and PCV13 serotypes)

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, MD PhD, Principal Investigator — University of the Witwatersrand, South Africa
Locations (1):
- Chris Hani Baragwanath Academic Hospital - DST/NRF VPD RMPRU, Soweto, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Olwagen CP, Izu A, Van der Merwe L, Jose L, Koen A, Madhi SA. Single priming and a booster dose of 10-valent and 13-valent pneumococcal conjugate vaccine (PCV) maintains suppression of vaccine serotype colonization in South African children at 3, 4, and 5 years of age: a single-centre, open-labelled, randomized trial. Expert Rev Vaccines. 2024 Jan-Dec;23(1):1011-1019. doi: 10.1080/14760584.2024.2417856. Epub 2024 Oct 22. PMID 39417218